CLINICAL TRIAL: NCT03222011
Title: Stricture Definition and Treatment (STRIDENT) Endoscopic Therapy Study
Acronym: STRIDENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Australasian Gastro Intestinal Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Kamm, Professor of Gastroenterology, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StVincentsMelbourneSTRIDENT2
Record Dates: First submitted 2017-07-06; First posted 2017-07-19 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Stricture; Bowel
Keywords: Crohn Disease; Inflammatory Bowel Disease; Intestinal stricture
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Constriction, Pathologic | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard endoscopic therapy (Active Comparator): Single endoscopic dilatation
  Interventions: Procedure: Standard (single) endoscopic stricture dilatation
- Intensive endoscopic therapy (Experimental): 3 endoscopic dilatations 3 weeks apart and possible needle knife strictureplasty
  Interventions: Procedure: Intensive endoscopic stricture dilatation

INTERVENTIONS:
Procedure: Standard (single) endoscopic stricture dilatation — single endoscopic stricture dilatation
  Arms: Standard endoscopic therapy
Procedure: Intensive endoscopic stricture dilatation — 3 endoscopic dilatations 3 weeks apart and possible needle knife strictureplasty
  Arms: Intensive endoscopic therapy

SUMMARY:
Two thirds of patients with Crohn's disease require intestinal surgery at some time in their life. Intestinal strictures, that is narrowing of the bowel due to inflammation and scarring, are the most common reason for surgery. Despite the high frequency, associated disability, and cost there are no are no treatment strategies that aim to improve the outcome of this disease complication. The STRIDENT (stricture definition and treatment) studies aim to develop such strategies.

DETAILED DESCRIPTION:
Prospective randomised controlled study. Patients with Crohn's Disease and symptomatic stricture(s) will undergo randomisation to receive standard or intensive endoscopic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease patients with intestinal stricture(s) identified on CT, MRI or endoscopy.

Exclusion Criteria:

* Acute bowel obstruction requiring urgent surgical intervention
* Deemed by treating physician to have high risk of acute bowel obstruction
* Concurrent active perianal sepsis
* Internal fistulising disease in association with strictures (entero-enteric stulas)
* Low rectal or anal strictures
* Evidence of dysplasia or malignancy from stricture biopsies or adjacent mucosal biopsies
* Patients for whom endoscopy is not suitable due to co-morbidities or clinical state
* Inability to give informed consent
* Suspected perforation of the gastrointestinal tract
* Pregnancy
* Inability to undergo MRI small bowel due to a contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in obstructive symptoms using the Obstructive Symptom Score (OSS). | 6 months
  The Obstructive Symptom Score (OSS) is a composite measure of the total number of days of obstructive abdominal pain and the severity over a fourteen-day period using a 5-point Likert scale. (no pain, mild, moderate, severe, unbearable)

SECONDARY OUTCOMES:
Improvement in obstructive symptoms using the Obstructive Symptom Score (OSS). | 3, 6 and 12 months
  The Obstructive Symptom Score (OSS) is a composite measure of the total number of days of obstructive abdominal pain and the severity over a fourteen-day period using a 5-point Likert scale. (no pain, mild, moderate, severe, unbearable)
Improvement in imaging parameters | 6 months
  MRI and intestinal ultrasound
Improvement in endoscopic features | 6 months
  Increased patency of strictures on endoscopy
Avoidance of surgery | 6 months
  Requirement for surgical resection of stricture
Improvement in patient reported outcomes (PROs) | 6 months
  IBDQ
Improvement in patient reported outcomes (PROs) | 6 months
  SF36
Technical success of procedure | At time of procedure
  Successful endoscopic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wright, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Bronte Holt, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne; Michael Kamm, MBBS PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schulberg JD, Hamilton AL, Wright EK, Holt BA, Sutherland TR, Ross AL, Vogrin S, Kamm MA. Repeated endoscopic dilation and needle-knife stricturotomy for Crohn's disease strictures. Gastrointest Endosc. 2025 Jan;101(1):202-206.e4. doi: 10.1016/j.gie.2024.09.031. Epub 2024 Sep 27. PMID 39343051